CLINICAL TRIAL: NCT05149144
Title: Comutti - A Research Project Dedicated to Finding Smart Ways of Using Technology for a Better Tomorrow for Everyone, Everywhere.
Acronym: COMUTTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Collaborators: Politecnico di Milano (Other); Massachusetts Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 868
Record Dates: First submitted 2021-11-25; First posted 2021-12-08 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Autism Spectrum Disorder
Keywords: non-verbal autistic children; minimally-verbal autistic children
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: audiosignal dataset creation and machine learning analysis (Experimental): Experimental: audiosignal dataset creation and processing; machine learning analysis, empirical evaluations
  Interventions: Diagnostic Test: Clinical evaluation of participants by means of Autism Diagnostic Observation Schedule; Behavioral: audio signal dataset creation and validation; machine learning analysis, empirical evaluations

INTERVENTIONS:
Diagnostic Test: Clinical evaluation of participants by means of Autism Diagnostic Observation Schedule — Clinical evaluation of participants by means of Autism Diagnostic Observation Schedule
Behavioral: audio signal dataset creation and validation; machine learning analysis, empirical evaluations — The project tests and adapts the technology developed at MIT for vocalization collection and labeling, and contributes to data gathering among Italian subjects (and their quality validation) in order to create a multi-cultural dataset and to enable cross-cultural studies and analyses. Next, the focus is placed on the analysis of harmonic features of the audio in the vocalizations of the dataset to identify recurring individual features and patterns corresponding to specific communications purposes or emotional states. Supervised and unsupervised machine learning approaches are developed and different machine learning algorithms will be compared to identify the most accurate ones for the project goal. Last, an exploratory evaluation of the vocalization-understanding machine learning model is conducted to test the usability and utility of the tool for vocalization interpretation.

SUMMARY:
According to World Health Organization, worldwide one in 160 children has an ASD. About around 25% to 30% of children are unable to use verbal language to communicate (non-verbal ASD) or are minimally verbal, i.e., use fewer than 10 words (mv-ASD). The ability to communicate is a crucial life skill, and difficulties with communication can have a range of negative consequences such as poorer quality of life and behavioural difficulties. Communication interventions generally aim to improve children's ability to communicate either through speech or by supplementing speech with other means (e.g., sign language, pictures, or AAC - Advanced Augmented Communication tools). Individuals with non- verbal ASD or mv-ASD often communicate with people through vocalizations that in some cases have a self-consistent phonetic association to concepts (e.g., "ba" to mean "bathroom") or are onomatopoeic expressions (e.g., "woof" to refer to a dog). In most cases vocalizations sound arbitrary; even if they vary in tone, pitch, and duration depending it is extremely difficult to interpret the intended message or the individual's emotional or physical state they would convey, creating a barrier between the persons with ASD and the rest of the world that originate stress and frustration. Only caregivers who have long term acquaintance with the subjects are able to decode such wordless sounds and assign them to unique meanings.

This project aims at defining algorithms, methods, and technologies to identify the communicative intent of vocal expressions generated by children with mv-ASD, and to create tools that help people who are not familiar with the subjects to understand these individuals during spontaneous conversations.

ELIGIBILITY:
Inclusion Criteria:

* having a clinical diagnosis of autism spectrum disorder according to DSM-5 criteria
* use fewer than 10 words

Exclusion Criteria:

* using any stimulant or non-stimulant medication affecting the central nervous system
* having an identified genetic disorder
* having vision or hearing problems
* suffering from chronic or acute medical illness

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Frequency of audio signal samples and their associated labels | immediately after the intervention
  Frequency (measured in number per hour) of audio signal samples (sounds and verbalizations) produced by each participant recorded during the hospital stays, in various contexts (i.e., during educational interventions and / or in moments of unstructured play) labeled as self-talk, delight, dysregulation, frustration, request, or social exchange.
  A small, wireless recorder (Sony TX800 Digital Voice Recorder TX Series) will be attached to the participant's clothing using strong magnets. Next, the adults (caregiver and / or operators) must associate the sounds produced by the child to an affective and / or to the probable meaning of the vocalization -labels- through the use of a web app.
Participant-specific harmonic features derived by the audio signal samples | immediately after the intervention
  Temporal and spectral audio features -i.e., pitch-related features, formants features, energy-related features, timing features, articulation features- extracted from the samples and used next for supervised and unsupervised machine learning analysis.
  The collected audio signal samples will be segmented in the proximity of the temporal locations of labels. Next, it will be segmented and associated with temporally adjacent labels (affective states or probable meaning of vocalizations). Audio harmonic features (temporal/phonetic characteristics) will be then identified for each participant using supervised/unsupervised machine learning analysis of audio signal samples. Through this process, participant-specific patterns corresponding to specific communications purposes or emotional states will be identified.
Accuracy of machine learning prediction | immediately after the intervention
  The classification accuracy of machine learning analysis, i.e., the number of correct predictions divided by the total number of predictions, which will be tested in a retained test set of recorded audio signal samples.
  This outcome measures will estimate the usability/utility of the developed tool for vocalization interpretion based on a machine learning analysis of the recorded audio signal samples.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Crippa, Ph.D., Principal Investigator — IRCCS Eugenio Medea
Locations (1):
- Scientific Institute, IRCCS Eugenio Medea, Bosisio Parini, Lecco, Italy

IPD SHARING:
Plan to Share IPD: No